CLINICAL TRIAL: NCT01234051
Title: Multicenter Phase II Study of Docetaxel and Oxaliplatin Combination in Patients With Locally Advanced or Metastatic Biliary Tract Cancer
Brief Title: Docetaxel and Oxaliplatin Combination With Locally Advanced or Metastatic Biliary Tract Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Korean South West Oncology Group (Network)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KSWOG 2010-1
Record Dates: First submitted 2010-10-28; First posted 2010-11-04 (Estimated); Last update posted 2011-12-12 (Estimated); Status verified 2010-11

CONDITIONS: Biliary Tract Cancer
MeSH Terms: conditions — Biliary Tract Neoplasms | interventions — Docetaxel; Oxaliplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Docetaxel, oxaliplatin, palliative chemotherapy (Experimental)
  Interventions: Drug: Docetaxel, Oxaliplatin

INTERVENTIONS:
Drug: Docetaxel, Oxaliplatin — 1. Treatment Schedule
  1.1. Docetaxel schedule Docetaxel 35 mg/m2 is administered on day 1 and day 8 by intravenously in 100 mL of 5% dextrose solution over 30 minutes. Dexamethasone 8mg is intravenously administered before 30 minutes, and then orally 4mg every 12 hours over 48 hours. In the event of a hypersensitivity reaction, dimethidine maleate, epinephrine, and intravenous fluids will be required.
  1.2. Oxaliplatin schedule Oxaliplatin 100 mg/m2 is given on day 1 by intravenous infusion in 500 mL of 5% dextrose solution over 120 minutes. Therapy will be repeated every 21 days.

SUMMARY:
1. Goals

   * The primary goal of this phase II trial is to:

   evaluate the response rate of combination chemotherapy with docetaxel and oxaliplatin in patients with locally advanced or metastatic BTC as first-line therapy

   Secondary goals are to:evaluate the treatment-related toxicities of this combination, investigate progression-free survival (PFS) and overall survival (OS) in this population
2. Design

The proposed clinical trial is an open label, non-comparative, multicenter phase II trial according to the two stage testing design by Simon.22

ELIGIBILITY:
Inclusion Criteria:

1. Patients who were diagnosed as adenocarcinoma of gallbladder or biliary tract histologically or cytologically
2. Unresectable locally advanced, metastatic, or recurrent biliary tract cancer
3. Patients must be ≥ 18 years old of age
4. ECOG performance status ≤ 2 (see Appendix C)
5. At least one lesion that can be measured by imaging (CT/MRI) according to the Response Evaluation Criteria in Solid Tumors (RECIST v1.1) (see Appendix D)
6. Estimated life expectancy of more than 3 months
7. Adequate bone marrow function (absolute neutrophil count [ANC] ≥ 1,500/µL, hemoglobin ≥ 9.0 g/dL [correction by transfusion is acceptable], and platelets ≥ 100,000/µL)
8. Adequate kidney function (serum creatinine < 1.5 x upper limit of normal [ULN])
9. Adequate liver function (serum total bilirubin < 3xULN; serum transaminases levels < 5xUNL)
10. Provision of fully informed consent prior to any study specific procedures

Exclusion Criteria:

1. Other tumor type than adenocarcinoma
2. Any previous history of chemotherapy for biliary tract cancer (prior neoadjuvant/adjuvant chemotherapy is allowed, if recurrence occurred more than 6 months after completion of previous chemotherapy)
3. Patients with second primary cancer (except, adequately treated non-melanoma skin cancer, curatively treated in-situ cancer of the cervix, or other solid tumors curatively treated with no evidence of disease for ≥5 years)
4. Patients who received radiotherapy on target lesion within 6 months prior to study treatment
5. Patients with defect of central nervous system (CNS) or any psychiatric disorders and CNS metastases
6. Patients who received major surgery within 4 weeks of starting study treatment or was not recovered from any effects of major surgery
7. Pregnant or breastfeeding women and women of childbearing potential not employing adequate contraception
8. Other serious illness or medical conditions A. Clinically significant cardiac disease (uncontrolled congestive heart disease despite treatment [NYHA class III or IV], symptomatic coronary artery disease, unstable angina or myocardial infarction, conduction abnormality like grade 2 AV block, serious arrhythmia needed for medication, uncontrolled hypertension) within 6 months prior to study entry B. Liver cirrhosis (≥ Child-Pugh class B) C. History of significant neurologic or psychiatric disorders including dementia or seizures D. Active uncontrolled infection E. Other serious underlying medical conditions which could impair the ability of the patient to participate in the study
9. Concomitant administration of any other experimental drug under investigation, or concomitant chemotherapy, hormonal therapy, or immunotherapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Estimated)
Dates: Start 2010-11; Primary Completion 2013-12 (Estimated); Study Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
Response rate | 2years

SECONDARY OUTCOMES:
Treatment-related toxicities | 2 years
  Number and proportion of patients with adverse events according to the NCI-CTCAE (v 4.0) as a measure of treatment-related toxicities
Progression free survival | 2 years
  Both survival curves will be calculated by Kaplan-Meier method and median value will be determined according to the survival curves.
  The median PFS and OS will be used for measure.
Overall survival | 2 years
  Both survival curves will be calculated by Kaplan-Meier method and median value will be determined according to the survival curves.
  The median PFS and OS will be used for measure.

CONTACTS AND LOCATIONS:
Overall Officials: Eun Ki Song, Principal Investigator — Chonbuk National Universitiy Hospital
Locations (1):
- Eun Ki Song, Chonbuk, South Korea